CLINICAL TRIAL: NCT05712330
Title: Exploratory Study of Respiratory Bacterial Infections or Superinfections and Colonizations in Patients With Spinal Muscular Atrophy Under NIV
Acronym: AVNIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0095
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Non Invasive Ventilation; Spinal Muscular Atrophy; Respiratory Bacterial Infection
Keywords: non invasive ventilation; Spinal Muscular Atrophy; Respiratory Bacterial Infection
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- non invasive ventilation (Experimental): SMA patients with NIV
  Interventions: Other: non invasive ventilation samples; Other: patient samples; Other: parent questionnaire

INTERVENTIONS:
Other: non invasive ventilation samples — machine samples for bacterial culture will be performed
Other: patient samples — Patient samples for sputum culture
Other: parent questionnaire — parent questionnaire

SUMMARY:
SMA (Spinal Muscular Atrophy) is a rare neuromuscular disease characterized by motoneuron damage. Symptoms consist of respiratory involvement with numerous respiratory infections and eventually respiratory failure, for which NIV (Non Invasive Ventilation) is often used. Ventilation machines are in close contact with the respiratory tract of patients. They contain heated water to humidify the circuit. These humid and warm environments are conducive to the development of bacteria such as Pseudomonas aeruginosa. In this context, it is interesting to look for the presence or absence of bacteria, in comparison with the respiratory ecology of the patients. The aim is to highlight the microbiological role of NIV on the occurrence of respiratory bacterial infections or secondary infections in patients with SMA. To do this, samples are taken from the machines, and ECBCs are performed on patients during respiratory physiotherapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AMS (previous diagnosis or new diagnosis during the inclusion period)
* Age from 0 to 12 years old
* Nusinersen treatment
* Benefiting from a NIV
* Current monitoring at the University Hospital of Amiens

Exclusion Criteria:

* Invasive ventilation on tracheotomy
* No ventilation
* Other treatment than Nusinersen or no treatment
* Parental refusal to participate in the study

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
number of hospitalization days for respiratory exacerbations with germs identical to protocol samples | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No